CLINICAL TRIAL: NCT01931241
Title: Phase I Randomized Placebo Controlled Double Blind SAD and MAD Study of Oral AHRO-001 to Assess Safety, Tolerability &PK in Volunteers w/Mild/Moderate Hypercholesteremia
Brief Title: Safety Study of Bile Acid to Treat Hypercholesteremia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AtheroNova Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHRO-001-12-101
Record Dates: First submitted 2013-07-10; First posted 2013-08-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hypercholesterolemia
Keywords: atherosclerosis; atherosclerotic heart disease; hypercholesteremia; atherosclerotic plaque; hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Coronary Artery Disease; Plaque, Atherosclerotic; Hyperlipidemias | interventions — hyodeoxycholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1, 500 mg (Experimental): Cohort 1 receives SDD 500 mg AHRO-001; one week later receives MDD of 500 mg bid 7 days, then 500 mg tid 7 days
  Interventions: Drug: AHRO-001
- Cohort 2, 750 mg (Experimental): Cohort 2 receives SD of 750 AHRO-001, then 7 days of 750 mg BID AHRO-001, then 7 days of 750 mg TID AHRO-001.
  Interventions: Drug: AHRO-001
- Cohort 3, 1000 mg (Experimental): Cohort 3 identical design as Cohorts 1 and 2, but SD is 1000 mg AHRO-001.
  Interventions: Drug: AHRO-001
- Cohort 4, 21 day dosing (Experimental): Cohort 4 receives 21 days tid administration of AHRO-001 using the best tolerated dose as determined by cohorts 1, 2 & 3
  Interventions: Drug: AHRO-001
- Cohort 5, 12 weeks dosing (Experimental): Cohort 5 receives 12 weeks tid administration of AHRO-001 using the best tolerated dose as determined by the first 4 cohorts.
  Interventions: Drug: AHRO-001

INTERVENTIONS:
Drug: AHRO-001 — Cohort 1: 500 mg/dose, given as a single dose then as bid x7days and tid x 7days Cohort 2: 750 mg/dose, given as a single dose then as bid x7days and tid x 7days Cohort 3: 1000 mg/dose, given as a single dose then as bid x7days and tid x7days Cohort 4: 21 days dosing given at best tolerated dose determined by cohorts 1-3 Cohort 5: 12 wks dosing given at best tolerated dose determined by cohorts 1-4
  Other Names: HDCA; Hyodeoxycholic acid

SUMMARY:
Preclinical data support the hypothesis that the administration of AHRO-001 reduces LDL cholesterol levels, improves HDL function, and finally, decreases atheromatous plaque burden.

DETAILED DESCRIPTION:
4 sequential dosing cohorts, each cohort beginning with single dose (SDD), single day exposure, followed by one week of multiple daily dosing (MDD) with bid exposure, a 4 day drug honeymoon, then one week of MDD utilizing tid exposure. Each subsequent cohort utilizes the same SDD/MDD design, starting with SDD higher than prior SDD but a SDD significantly lower than prior tid MDD cohort just completed, the overall goal being to provide gradually increasing dose exposure contingent on satisfactory safety and tolerability of lower doses in the previous groups. Cohort 4 (MDD) utilizes best dose determined by Cohorts 1, 2 & 3 for 21 days.

Estimated Duration of Subject Participation: 8-9 weeks

Under Protocol Amendment Version 5.0, an additional cohort, Cohort 5, will concomitantly enroll 48 volunteers randomized to receive either AHRO-001 or placebo. Volunteers included in the study may be either currently receiving or not receiving a statin treatment. The 48 volunteers in Cohort 5 will thus be allocated to 3 treatment groups with 16 volunteers enrolled per group:

Group A: AHRO-001 alone Group B: Statin + AHRO-001 Group C: Placebo

SUBJECT POPULATION:

Healthy volunteers, both males & infertile females, with asymptomatic mild to moderate hypercholesterolemia

ELIGIBILITY:
Key Inclusion Criteria:

* Males OR infertile Females
* 18-70 years of age, inclusive
* Asymptomatic mild to moderate hypercholesterolemia, (LDL =110-220 mg/dL)
* Cohort 5: on no statin or on a stable statin dose not meeting LDL >110 mg%

Key Exclusion criteria

* Fasting triglycerides <90 or >250 mg/dl (<0.85 mmol/l or >2.8 mmol/l)
* Body Mass Index (BMI) <18 or >34 kg/m2
* Diabetes mellitus (FBS > 125 mg% (>6.94 mmol/l)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >ULN
* Serum creatinine >ULN for gender
* Hemoglobin <11.5 g/dL
* Female volunteers of childbearing potential
* History of cancer in past 5 years
* Any disease requiring medication
* Use of investigational medication in past 3 months
* Positive results for illegal drugs, HBsAg, HBsAb, HCV or HIV
* Cohort 5:Prescription lipid lowering medications other than a statin in past 4 wks
* Cohort 5: History of gastrointestinal tract surgical resection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Participants will be followed through the course of their participation, approximately 8 weeks
  To assess the safety, tolerability and pharmacokinetics of AHRO-001 when administered first as a single daily dose x 1 day, then by a graduated increase from daily dosing x 1day to twice daily dosing x7 days, and ultimately to thrice daily dosing x7. Next dose can be started as soon as 6 volunteers will finish 2 weeks of administration of the previous dose. All dose increases occur only after drug washout and are only undertaken after medical review of the previous dose as determined by symptoms, vital signs, clinical examination, clinical laboratory results, urinalyses, electrocardiograms and adverse event reporting declares that progression of dosing is safe and appropriate

SECONDARY OUTCOMES:
Number of participants with adverse events | Participants will be followed through the course of their participation, approximately 8 weeks
  To assess the safety, tolerability and pharmacokinetics of AHRO-001 dosed tid for 21 days at best tolerated dose as determined in Cohorts 1-3.
Number of participants with adverse effects | Participants will be followed through the course of their participation, approximately 16 weeks
  To assess the safety, tolerability and pharmacokinetics of AHRO-001 administered orally as a tid regimen for 12 weeks in the presence or absence of a statin, at a dose determined by safety in the first 4 dose cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K. Wedel, MD, Study Chair — AtheroNova CMO
Locations (1):
- City Hospital #15, Moscow, Russia